CLINICAL TRIAL: NCT03212521
Title: A Single Arm, Open Label, Multicenter Study to Evaluate the Efficacy and Safety of Glecaprevir (GLE)/Pibrentasvir (PIB) in Treatment Naïve Adults With Chronic Hepatitis C Virus (HCV) Genotypes 1 - 6 Infection and Aspartate Aminotransferase to Platelet Ratio Index (APRI) ≤ 1
Brief Title: Efficacy and Safety of 8-weeks of Glecaprevir/Pibrentasvir in Treatment-Naïve Adults With HCV Genotype 1-6 and Aspartate Aminotransferase to Platelet Ratio Index (APRI) ≤1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-133; 2016-004876-23 (EudraCT Number)
Expanded Access: NCT03123965 (Approved for marketing)
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: chronic hepatitis C virus (HCV); Hepatitis; HCV genotype; aspartate aminotransferase; platelet; Aspartate aminotransferase to Platelet Ratio Index (APRI); glecaprevir; pibrentasvir; Sustained Virologic Response 12 weeks post dosing (SVR12)
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Hepatitis | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Glecaprevir/Pibrentasvir (Experimental): Participants received oral glecaprevir/pibrentasvir (300 mg/120 mg) once daily with food for 8 weeks.
  Interventions: Drug: Glecaprevir/Pibrentasvir

INTERVENTIONS:
Drug: Glecaprevir/Pibrentasvir — Glecaprevir/pibrentasvir 100 mg/40 mg co-formulated tablets taken orally as 3 tablets once a day.
  Other Names: ABT-493/ABT-530; MAVYRET™

SUMMARY:
A study to evaluate the efficacy and safety of glecaprevir(GLE)/pibrentasvir(PIB) in treatment-naïve participants with chronic hepatitis C virus (HCV) genotypes 1-6 infection and with an aspartate aminotransferase to platelet ratio index (APRI) of less than or equal to 1.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C virus (HCV) genotype (GT) 1, 2, 3, 4, 5, or 6 infection. Mixed GT and indeterminate GT may be acceptable.
* Aspartate aminotransferase (AST) to platelet ratio index (APRI) score of less than or equal to 1, at time of screening.
* Does not have current active hepatitis B virus infection defined as:

  * positive hepatitis B surface antigen (HBsAg), OR
  * hepatitis B virus (HBV) deoxyribonucleic acid (DNA) > lower limit of quantification (LLOQ) in subjects with isolated positive anti-hepatitis B core (HBc) (i.e., negative HBsAg and anti-hepatitis B surface[HBs])
* Platelets ≥ 150,000 cells/mm³
* Albumin ≥ lower limit of normal (LLN)
* Positive anti-HCV antibody (Ab) AND plasma HCV ribonucleic acid (RNA) viral load ≥ 1,000 IU/mL at Screening and for at least 6 months before Screening.
* No past history/evidence of cirrhosis.
* No history of hepatocellular carcinoma.
* Hepatitis C virus treatment-naïve (had not received a single dose of any approved or investigational anti-HCV medication).
* If female, the subject must not be pregnant, breastfeeding, or considering becoming pregnant during the study and for 30 days after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (42):
- United States (11):
  - Parkway Medical Center /ID# 161261, Birmingham, Alabama
  - Arkansas Gastroenterology /ID# 161266, North Little Rock, Arkansas
  - UC Davis Medical Center /ID# 161138, Sacramento, California
  - Yale University /ID# 161258, New Haven, Connecticut
  - Univ Maryland School Medicine /ID# 161157, Baltimore, Maryland
  - Digestive Disease Associates - Baltimore /ID# 161260, Baltimore, Maryland
  - University of Michigan Hospitals /ID# 161265, Ann Arbor, Michigan
  - Northwest Gastroenterology Cli /ID# 161257, Portland, Oregon
  - Liver Associates of Texas, P.A /ID# 161262, Houston, Texas
  - University of Vermont Medical Center /ID# 161263, Burlington, Vermont
  - Digestive and Liver Disease Sp /ID# 161259, Norfolk, Virginia
- Bulgaria (2):
  - DCC Aleksandrovska /ID# 161340, София, Sofia
  - DCC Mladost M /ID# 161339, Varna
- Canada (4):
  - South Health Campus /ID# 161385, Calgary, Alberta
  - The Moncton Hospital /ID# 161384, Moncton, New Brunswick
  - Brampton Civic Hospital /ID# 161380, Brampton, Ontario
  - Toronto Liver Centre /ID# 161381, Toronto, Ontario
- France (4):
  - Hopital Saint Joseph /ID# 161571, Marseille, Bouches-du-Rhone
  - CHU de Rennes - PONTCHAILLOU /ID# 161492, Rennes, Brittany Region
  - CHU de Besancon - Jean Minjoz /ID# 161485, Besançon, Doubs
  - Hopitaux de Brabois Adultes /ID# 161482, Vandœuvre-lès-Nancy, Lorraine
- Germany (4):
  - Universitätsklinikum Frankfurt /ID# 161397, Frankfurt am Main, Hesse
  - Universitaetsmedizin der Johannes-Gutenberg Universität Mainz /ID# 161396, Mainz, Rhineland-Palatinate
  - Charité Universitätsmedizin Campus Mitte /ID# 161395, Berlin
  - ICH Study Center GmbH & Co KG /ID# 161394, Hamburg
- Poland (4):
  - Centrum Badan Klinicznych /Id# 162218, Wroclaw, Lower Silesian Voivodeship
  - HepID - Diagnostyka I Terapia /ID# 162219, Lublin, Lublin Voivodeship
  - Uniwersytecki Szpital Kliniczn /ID# 162216, Bialystok
  - ID Clinic /ID# 162217, Mysłowice
- Innovative Care P.S.C. /ID# 162787, San Juan, Puerto Rico
- Russia (3):
  - A. F. Agafonov Republican Clin /ID# 163164, Kazan', Tatarstan, Respublika
  - South Ural State Medical univ /ID# 163163, Chelyabinsk
  - A.I. Evdokimov Moscow State Un /ID# 163162, Moscow
- Spain (5):
  - Hospital Fundacion Alcorcon /ID# 161436, Alcorcón
  - Hospital Clinic de Barcelona /ID# 161437, Barcelona
  - Hospital Vall d'Hebron /ID# 162022, Barcelona
  - Hosp Uni Virgen de la Victoria /ID# 164383, Málaga
  - Complexo Hospitalario universi /ID# 165603, Pontevedra
- United Kingdom (4):
  - Bradford Teaching Hospitals /ID# 161424, Bradford
  - Glasgow Royal Infirmary /ID# 161458, Glasgow
  - Gloucester Royal Hospital /ID# 161423, Gloucester
  - Freeman Hospital /ID# 161459, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Fontana RJ, Lens S, McPherson S, Elkhashab M, Ankoma-Sey V, Bondin M, Dos Santos AGP, Xue Z, Trinh R, Porcalla A, Zeuzem S. Efficacy and Safety of 8 Weeks of Glecaprevir/Pibrentasvir in Treatment-Naive, HCV-Infected Patients with APRI </= 1 in a Single-Arm, Open-Label, Multicenter Study. Adv Ther. 2019 Dec;36(12):3458-3470. doi: 10.1007/s12325-019-01123-0. Epub 2019 Oct 23. PMID 31646465

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 40 sites in Bulgaria, Canada, France, Germany, Poland, Russian Federation, Spain, United Kingdom, and the United States (including Puerto Rico).
Period: Overall Study
Arm/Group | Glecaprevir/Pibrentasvir
Started | 230
Completed | 223
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 230
Age, Continuous [Median (Full Range); unit: years] | 48 [19 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25
  Not Hispanic or Latino | 205
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 207
  Black or African American | 13
  Asian | 10
Hepatitis C Virus (HCV) Genotype [Count of Participants; unit: Participants]
  Genotype 1 | 151
  Genotype 2 | 33
  Genotype 3 | 35
  Genotype 4 | 9
  Genotype 5 | 0
  Genotype 6 | 2
Aminotransferase/Platelet Ratio Index (APRI) [Median (Full Range); unit: ratio] — APRI is used to determine the likelihood of hepatic fibrosis and cirrhosis in patients with hepatitis C. APRI is calculated from the level of aspartate aminotransferase (AST) measured in a blood test (international units per liter [IU/L)] and platelet count (platelets/cubic millimeter) according to the following formula:
  APRI = [(AST/upper limit of the normal range (ULN) of AST) x 100] / Platelet count
  APRI scores of less than or equal to 1 have a good performance characteristic for excluding the presence of cirrhosis.
  ratio | 0.41 [0.13 to 1.00]
HCV Ribonucleic Acid (RNA) Concentration [Median (Full Range); unit: Log₁₀ IU/mL] | 6.29 [2.22 to 7.74]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in the Modified Intention-to-Treat Population With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification (LLOQ; 15 IU/mL) 12 weeks after the last dose of study drug.
  The 95% confidence interval (95%CI) was calculated using the Wilson's score method.
  Efficacy was to be established if the lower bound of the 95%CI was greater than the threshold of 92.4%, based on the historical rate observed in glecaprevir/pibrentasvir registrational studies in treatment-naïve, non-cirrhotic patients (98.4%) minus a margin of 6%.
Time Frame: 12 weeks after the last actual dose of study drug, Week 20
Population: The modified intention-to-treat (mITT) population includes all enrolled participants who received at least 1 dose of study drug, excluding participants who did not achieve SVR12 for reasons other than virologic failure, such as missing SVR12 data (5 participants) or premature study drug discontinuation (3 participants).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 222
percentage of participants | 100.0 [98.3 to 100.0]

2. Secondary Outcome: Percentage of Participants in the Intention-to-Treat Population With SVR12
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the LLOQ (15 IU/mL) 12 weeks after the last dose of study drug.
  The 95% confidence interval was calculated using the normal approximation to the binomial distribution. Efficacy was to be established if the lower bound of the 95%CI was greater than the threshold of 91.4%, based on the mITT threshold minus an expected 1% rate of non-virological SVR failures.
Time Frame: 12 weeks after the last actual dose of study drug, Week 20
Population: The intention-to-treat (ITT) population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 230
percentage of participants | 96.5 [94.2 to 98.9]

3. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as one of the following conditions:
  * confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < 15 IU/mL during the Treatment Period; or
  * confirmed increase from nadir in HCV RNA (two consecutive HCV RNA measurements > 1 log₁₀ IU/mL above nadir) at any time point during the Treatment Period; or
  * HCV RNA ≥ 15 IU/mL at end of treatment with at least 6 weeks of treatment, where the HCV RNA value must be collected on or after Study Drug Day 36 and study drug duration ≥ 36 days.
Time Frame: Up to 8 weeks
Population: Intention-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 230
percentage of participants | 0.0 [0.0 to 1.6]

4. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment.
Time Frame: From the end of treatment (Week 8) through 12 weeks after the last dose of study drug (Week 20)
Population: Intention-to-treat population with HCV RNA < 15 IU/mL at the end of treatment, at least one post-treatment HCV RNA value, and who completed the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 225
percentage of participants | 0.0 [0.0 to 1.7]

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after the last dose of study drug; 12 weeks
Arm/Group | Glecaprevir/Pibrentasvir
All-Cause Mortality (participants affected / at risk) | 0/230
Serious Adverse Events (participants affected / at risk) | 4/230
Other Adverse Events (participants affected / at risk) | 46/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glecaprevir/Pibrentasvir (N=230)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (1)
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 1 (1)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glecaprevir/Pibrentasvir (N=230)
FATIGUE (General disorders) | 17 (17)
HEADACHE (Nervous system disorders) | 29 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT03212521/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT03212521/SAP_001.pdf